CLINICAL TRIAL: NCT05977413
Title: NOTIFY-OUTCOMES (New Observations Taking Information From Yesterday)
Brief Title: NOTIFY (New Observations Taking Information From Yesterday)
Acronym: NOTIFY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was never started because it was not funded.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Maron, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 71202
Record Dates: First submitted 2023-07-19; First posted 2023-08-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-Clinician CAC Notification (Experimental): The CAC Notification intervention sent to both patients and clinicians has five features. 1) Results of a high CAC score (>100 AU) detected on the patient's prior chest CT, 2) an image of the patient's CAC clearly marked, 3) a recommendation to have a patient-clinician risk discussion, 4) specific statin dosing recommended by guidelines, and 5) a link to the prevention gidelines.
  Interventions: Other: CAC Notification
- Clinician Guideline Reminder (Other): The Guideline Reminder intervention sent to primary care clinicians has five features. 1) A reminder that all patients should have their 10-year risk for ASCVD events calculated, 2) a figure of the recommended treatment algorithm according to ASCVD 10-year risk, 3) a nudge that patients who qualify for lung cancer screening are generally at high ASCVD risk, 4) a reminder that patients at elevated risk should be engaged in shared decision-making to discuss statin therapy and other preventive interventions, and 5) access to the complete ACC/AHA Primary Prevention Guidelines and the online 10-year ASCVD risk estimator.
  Interventions: Other: Clinician Guideline Reminder

INTERVENTIONS:
Other: CAC Notification — Patient-Clinician CAC Notification. The CAC Notification intervention sent to both patients and clinicians has five features. 1) Results of a high CAC score (>100 AU) detected on the patient's prior chest CT, 2) an image of the patient's CAC clearly marked, 3) a recommendation to have a patient-clinician risk discussion, 4) specific statin dosing recommended by guidelines, and 5) a link to the prevention gidelines.
  Arms: Patient-Clinician CAC Notification
Other: Clinician Guideline Reminder — The Guideline Reminder intervention sent to primary care clinicians has five features. 1) A reminder that all patients should have their 10-year risk for ASCVD events calculated, 2) a figure of the recommended treatment algorithm according to ASCVD 10-year risk, 3) a nudge that patients who qualify for lung cancer screening are generally at high ASCVD risk, 4) a reminder that patients at elevated risk should be engaged in shared decision-making to discuss statin therapy and other preventive interventions, and 5) access to the complete ACC/AHA Primary Prevention Guidelines and the online 10-year ASCVD risk estimator.
  Arms: Clinician Guideline Reminder

SUMMARY:
This trial will investigate whether notifying patients and their clinicians of the presence of moderate or severe coronary artery calcium on a low-dose CT scan performed for lung cancer screening results in a lower incidence of death, nonfatal myocardial infarction, or nonfatal stroke as compared with practice guideline reminders.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* No known ASCVD
* Lung cancer screenee with low dose CT scan (LDCT) within the last 5 years
* Coronary artery calcium (CAC) score on LDCT >100 Agatston units (AU)
* Not taking a statin or other lipid-lowering therapy (e.g., ezetimibe, bempedoic acid, or PCSK9-lowering therapy)

Exclusion Criteria:

* Dementia or other neuropsychiatric disorder that interferes with medication adherence
* CAC scan, coronary CT angiogram, or invasive angiogram since LDCT
* Statin medication intolerance or allergy
* Life expectancy <2 years, e.g., metastatic cancer or active cancer undergoing chemotherapy

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2032-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of death, nonfatal myocardial infarction, or nonfatal stroke | 6 years

SECONDARY OUTCOMES:
Rate of All-cause Death | 6 years
  Number (%) of participants in each treatment group with death from any cause.
Rate of Cardiovascular Death | 6 years
  Number (%) of participants in each treatment group with cardiovascular death
Rate of Nonfatal Myocardial Infarction | 6 years
  Number (%) of participants in each treatment group with nonfatal myocardial infarction
Rate of Nonfatal Stroke | 6 years
  Number (%) of participants in each treatment group with nonfatal stroke
Initial lipid-lowering therapy prescription rate | within 6 months of 1st notification
  Number (%) of participants in each treatment group with active prescriptions of lipid-lowering therapy at 6 months following randomization
Number of Participants with active lipid-lowering therapy prescriptions | At 18 months
  Persistence of need for lipid-lowering therapy at 18 months following randomization.
Number of revascularization procedures (PCI, CABG, carotid artery revascularization, or peripheral artery revascularization) | 6 years
  Number of revascularization procedures (PCI, CABG, carotid artery revascularization, or peripheral artery revascularization)

OTHER OUTCOMES:
Rate of Specific Statin Prescribed and Statin Dose | 1 year post randomization
  Rate of prescription of specific statins at specific doses
Rate of Prescription of Non-statin Lipid-lowering Medications | 1 year post randomization
  Rate of prescription of specific non-statins
Rate of Aspirin Prescription | 1 year post randomization
  Rate of aspirin prescription by treatment group
Number of Antihypertensive Medications | 1 year post randomization
  Number of antihypertensive medications prescribed per participant by treatment group
Median LDL-C Concentration | 1 year post randomization
  Median LDL cholesterol concentration by treatment group
Percentage of participants with LDL-C <70 mg/dL | 1 year post randomization
  Percentage of participants with LDL-C <70 mg/dL by treatment group
Systolic blood pressure | 1 year post randomization
  Median systolic blood pressure value in mmHg by treatment group
Percentage of participants with Systolic Blood Pressure <130 mmHg | 1 year post randomization
  Percentage of participants with systolic blood pressure <130 mmHg by treatment group
Body Mass Index | 1 year post randomization
  Median body mass index value by treatment group
Total number of primary care clinical encounters during the trial | 6 years
Number of cardiology encounters | 6 years
Number of cardiovascular diagnostic noninvasive tests | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: David J Maron, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandhu AT, Rodriguez F, Ngo S, Patel BN, Mastrodicasa D, Eng D, Khandwala N, Balla S, Sousa D, Maron DJ. Incidental Coronary Artery Calcium: Opportunistic Screening of Previous Nongated Chest Computed Tomography Scans to Improve Statin Rates (NOTIFY-1 Project). Circulation. 2023 Feb 28;147(9):703-714. doi: 10.1161/CIRCULATIONAHA.122.062746. Epub 2022 Nov 7. PMID 36342823
- [Background] Eng D, Chute C, Khandwala N, Rajpurkar P, Long J, Shleifer S, Khalaf MH, Sandhu AT, Rodriguez F, Maron DJ, Seyyedi S, Marin D, Golub I, Budoff M, Kitamura F, Takahashi MS, Filice RW, Shah R, Mongan J, Kallianos K, Langlotz CP, Lungren MP, Ng AY, Patel BN. Automated coronary calcium scoring using deep learning with multicenter external validation. NPJ Digit Med. 2021 Jun 1;4(1):88. doi: 10.1038/s41746-021-00460-1. PMID 34075194